CLINICAL TRIAL: NCT03870360
Title: Health Promotion in the Prevention of Anxiety and Depression: the Happy Older Latinos Are Active (HOLA Study)
Brief Title: Preventing Anxiety and Depression in Older Hispanics
Acronym: HOLAA&D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daniel Enrique Jimenez, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20180816; R01MD012610 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOLA: A Culturally-Tailored Health Promotion Intervention (Experimental): 16 week, multicomponent, health promotion intervention
  Interventions: Behavioral: HOLA Component 1; Behavioral: HOLA Component 2; Behavioral: HOLA Component 3; Behavioral: HOLA Component 4
- Healthy lifestyles education program (Active Comparator): Educational material on mental health, physical activity, and information on community resources
  Interventions: Behavioral: Healthy lifestyles education program

INTERVENTIONS:
Behavioral: HOLA Component 1 — At week 1 and week 8 participants will meet individually with Community Health Worker (CHW) for 30 minutes for a manualized social and physical activation session.
  Arms: HOLA: A Culturally-Tailored Health Promotion Intervention
Behavioral: HOLA Component 2 — A CHW led 45 minute (10 minutes of stretching and warm up, followed by 30 minutes of walking with a 5 minute cool down) group walk session of six participants at a time done 3 times a week that utilized interval training that slowly gradually increases in intensity.
  Arms: HOLA: A Culturally-Tailored Health Promotion Intervention
Behavioral: HOLA Component 3 — A CHW led pleasant event discussion, asking each participant to identify a pleasant event. This task is done in conjunction with the cool down of HOLA 2.
  Arms: HOLA: A Culturally-Tailored Health Promotion Intervention
Behavioral: HOLA Component 4 — One booster walking session twice a month for six months post intervention for reinforcement, then one booster walking session a month for eighteen months.
  Arms: HOLA: A Culturally-Tailored Health Promotion Intervention
Behavioral: Healthy lifestyles education program — Biweekly telephone check in calls for the first 16 weeks followed by monthly check in calls during the two year follow up period.
  Arms: Healthy lifestyles education program

SUMMARY:
The purpose of this study is to look at the best ways to prevent anxiety and depression in older Latino adults who are at risk for developing anxiety and depression. Participants will be randomized to either a health promotion intervention or a healthy lifestyles education program.

DETAILED DESCRIPTION:
Given the prevalence and morbidity of depression in later life, the inadequacies of current treatment approaches for averting years living with disability, the inequities in access to the mental health care delivery system, and the workforce shortages to meet the mental health needs of older Latinos, development and testing of innovative strategies to prevent depression and anxiety are of great public health significance and have the potential to change practice.

ELIGIBILITY:
Inclusion Criteria:

* Latino (self-identified);
* Age 60+;
* Subthreshold depression defined as a score ≥ 5 on the Patient Health Questionnaire (PHQ-9), OR subthreshold anxiety as defined as a score ≥ 5 on the GAD-7;
* Do not meet criteria for current MDD or GAD as indicated by the Mini International Neuropsychiatric Inventory (MINI);
* Voluntary informed consent for participation in the study by the participant or by the participant's legally designated guardian or conservator;
* Medical clearance for participation in a health promotion intervention by a physician, physician's assistant, or nurse practitioner;
* Not taking steroidal or anti-inflammatory medication (including NSAIDs) within 2 weeks of treatment randomization;
* Expect to be resident in Miami for the subsequent 2 years.

Exclusion Criteria:

* Have met criteria for major depressive disorder or generalized anxiety disorder within the past 12 months;
* Have met criteria for alcohol or other substance abuse disorders within the past 12 months;
* Are currently receiving antidepressant medication or participating in other mental health treatment;
* Have a lifetime history of bipolar disorder or other psychotic disorder including major depression with psychotic features;
* Have a diagnosis of any neurodegenerative disorder or dementia (Parkinson's disease, Alzheimer's, vascular, frontotemporal dementia, etc.) or significant cognitive impairment as indicated by a Mini Mental Status Exam (MMSE) score <24;
* Are current tobacco smokers since smoking influences systemic inflammation;
* Have contraindications to physical activity outlined in the American College of Sports Medicine standards;
* Have high suicide risk, i.e., intent or plan to attempt suicide in the near future (a response of "yes" to questions 3, 4, and/or 5 on the Paykel Questionnaire;
* Are unable to complete 10 m walk test;
* Currently residing in a nursing or group home;
* Have a terminal physical illness expected to result in the death within one year;
* Any evidence of current infection; and
* Have an acute or severe medical illness that precludes them from safely participating in a health promotion intervention (further defined in the protocol).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in risk factors for major depressive disorder (MDD) | Baseline, 16 weeks, 6, 12, 18, and 24 months
  As measured by the Beck Depression Inventory that has a range of scores from 0-63 with scores of 0-9 being minimal depression, 10-18 mild depression, 19-29 moderate depression, and 30-63 severe depression.
Change in risk factors for generalized anxiety disorder (GAD) | Baseline, 16 weeks, 6, 12, 18, and 24 months
  As measured by the Beck Anxiety Inventory that has a range of scores from 0-63 with scores 0-21 low anxiety, 22-35 moderate anxiety, and 36+ potentially concerning levels
Incidence of generalized anxiety disorder | 2 years
  As measured by the Structured Clinical Interview for the Diagnostic and Statistical Manual 5th edition (SCID-5), a structured clinical interview used for diagnosis.
Recurrence of generalized anxiety disorder | 2 years
  As measured by the SCID-5, a structured clinical interview used for diagnosis.
Incidence of major depression disorder | 2 years
  As measured by the SCID-5, a structured clinical interview used for diagnosis.
Recurrence of major depression disorder | 2 years
  As measured by the SCID-5, a structured clinical interview used for diagnosis.

SECONDARY OUTCOMES:
Change in pro-inflammatory markers | Baseline, 16 weeks, 12, and 24 months
  Obtained from plasma samples
Change in anti-inflammatory markers | Baseline, 16 weeks, 12, and 24 months
  Obtained from plasma samples
Change in physical functioning as measured by the physical performance battery | Baseline, 16 weeks, 6, 12, 18, and 24 months
  The battery assesses static balance, leg strength, normal gait speed, and narrow walk for dynamic balance using the 6-minute walk test, the timed up and go test, and the gallon jug shelf transfer test.
Change in quality of life | Baseline, 16 weeks, 6, 12, 18, and 24 months
  As measured by the Short Form Health Survey 12 (SF-12). The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). MCS scores range from 0 to 100, higher scores indicate better mental health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Jimenez, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No